CLINICAL TRIAL: NCT07070011
Title: Small Extracellular Vesicle miRNAs as Predictive Biomarkers for Immunochemotherapy Efficacy in Extensive-stage Small Cell Lung Cancer
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital of Shanghai Jiao Tong University (Other)
Responsible Party: Principal Investigator, Wei Zhang, Chief Physician, Shanghai Chest Hospital of Shanghai Jiao Tong University
Other Study IDs: IS2109-(LGZ)
Record Dates: First submitted 2025-06-02; First posted 2025-07-17 (Actual); Last update posted 2025-07-17 (Actual); Status verified 2025-07

CONDITIONS: Extensive-stage Small Cell Lung Cancer (ES-SCLC)
Keywords: small cell lung cancer; immunochemotherapy; sEV miRNAs; predictive biomarkers
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 38 Days
Biospecimen Retention: Samples Without DNA — Blood samples from patients with small cell lung cancer before receiving immunotherapy combined with chemotherapy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Partial Response (PR), Stable Disease (SD) and Progressive Disease (PD).: Partial Response (PR): Defined as a reduction in the sum of the diameters of target lesions by ≥30% from baseline, in the absence of new lesions. This indicates effective treatment with significant tumor shrinkage.
  Stable Disease (SD): Defined as neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for Progressive Disease (i.e., the sum of the diameters of target lesions shows a change ranging from a decrease of <30% to an increase of <20%), in the absence of new lesions. This indicates that the disease has not worsened, but a significant reduction in tumor burden has not been achieved.
  Progressive Disease (PD): Defined as an increase in the sum of the diameters of target lesions by ≥20% (taking as reference the smallest sum on study), and/or the appearance of one or more new lesions. This signifies treatment failure, necessitating a modification of the therapeutic regimen.
  Interventions: Combination Product: EC/EP + ICIs

INTERVENTIONS:
Combination Product: EC/EP + ICIs — Collect blood samples from patients with small cell lung cancer before receiving immunotherapy combined with chemotherapy.

SUMMARY:
This study aims to investigate the clinical value of small extracellular vesicle (sEV) miRNAs as predictive biomarkers for immunochemotherapy efficacy in extensive-stage small cell lung cancer (ES-SCLC). ES-SCLC represents a highly aggressive neuroendocrine malignancy, where the current standard first-line treatment combining immune checkpoint inhibitors with chemotherapy lacks predictive biomarkers for individualized therapeutic strategies.

A prospective observational cohort will be established at Shanghai Chest Hospital, enrolling treatment-naïve ES-SCLC patients. Distinct miRNA signatures differentiating responders from non-responders will be identified through pretreatment serum sEV miRNA sequencing and differential expression analysis. These findings may provide novel liquid biopsy biomarkers to guide personalized treatment strategies and optimize clinical decision-making in ES-SCLC management.

ELIGIBILITY:
Inclusion Criteria:

Requirements for patients enrolled in the project:

1. The pathological diagnosis of the patient is ESSCLC;
2. ECOG score 0 or 1；
3. The patient is receiving immunotherapy combined with chemotherapy for the first time and has no history of chemotherapy treatment;
4. Patients with complete clinical sample information who meet the inclusion requirements

Exclusion Criteria:

1. Patients whose pathological diagnosis does not meet the requirements;
2. Patients whose ECOG staging does not meet the requirements;
3. Patients with a history of chemotherapy, immunotherapy, or immunotherapy combined with chemotherapy;
4. Patients with incomplete clinical sample information and follow-up information;

Ages: 45 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: ES-SCLC (extensive-stage small cell lung cancer) patients with an ECOG performance status of 0-1 and no prior exposure to immunotherapy or chemotherapy.
Sampling Method: Non-Probability Sample
Enrollment: 38 (Estimated)
Dates: Start 2023-01-03 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Tumor Response Status per RECIST 1.1 | 6 to 8 weeks
  * Assessment Tool: RECIST 1.1 criteria ;
  * Unit of Measure: Number of patients (n) and percentage (%) ;
  * Data Aggregation Method: Calculation of proportions of patients in each response category (PR/SD/PD);
  Definitions:
  * Partial Response (PR): ≥30% reduction in the sum of diameters of target lesions from baseline (absence of new lesions) ;
  * Stable Disease (SD): Change in the sum of diameters ranging from <30% reduction to <20% increase (absence of new lesions) ;
  * Progressive Disease (PD): ≥20% increase in the sum of diameters (reference: smallest sum recorded) and/or appearance of new lesions ;
Baseline Serum sEV miRNA Expression Levels | Baseline (pre-treatment)
  * Measurement Tool: Next-generation sequencing (NGS) ;
  * Unit of Measure: Standardized expression values (CPM, Counts Per Million) ;
  * Data Aggregation Method: Descriptive statistics (mean ± SD or median [IQR]) of expression levels by response groups ;
  * Procedure:
    1. Pre-treatment serum collection ;
    2. sEV isolation ;
    3. miRNA extraction ;
    4. NGS sequencing ;
    5. Bioinformatic normalization (CPM) .

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No